CLINICAL TRIAL: NCT03810248
Title: Association Between Obstructive Sleep Apnea and Bruxism: A Retrospective Study
Brief Title: Association Between Obstructive Sleep Apnea and Bruxism
Status: Completed | Type: Observational
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Noéli Boscato, PhD, Associate Professor, Federal University of Pelotas
Other Study IDs: FUPelotas 4
Record Dates: First submitted 2018-11-06; First posted 2019-01-18 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Bruxism, Sleep; Obstructive Sleep Apnea
Keywords: sleep bruxism; polisomnography
MeSH Terms: conditions — Sleep Bruxism; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this retrospective observational study will be to investigate the between the Obstructive Sleep Apnea Syndrome (OSAS) and Sleep Bruxism (SB), in individuals diagnosed through polysomnography (PSG).

DETAILED DESCRIPTION:
The SB and OSAS are sleep disorders with great importance for dentistry. The OSAS is characterized by partial or total obstruction of the upper airways. SB is defined as a repetitive activity of the mandibular musculature characterized by the tightening or grinding of the teeth and/or by the retrusion or propulsion of the mandible. This study retrospective observational will be evaluation to investigate the association between OSAS and SB. Data from PSG and medical records (n=640) will be collected from January 2012 to July 2018 at "Instituto do Sono de Pelotas (ISP)".

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 20 to 60 years) and elderly (aged > 60 years) (WHO-World Health Organization, 2015) who was undergone PSG at the "Instituto do Sono de Pelotas (ISP)";
* Have completed all the respective PSG reports.

Exclusion Criteria:

•Those which the participants were unable to answer the questionnaires and who presented a history of epilepsy that could interfere in the results of PSG.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals who have undergone polysomnography at the Instituto do Sono de Pelotas (ISP) between March 2012 and July 2018, who meet inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 640 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Tabulation of polysomnographic report related to sleep efficiency | The deadline is until May 2020 to have all data collected
  These data are provided from the medical report generated in the polysomnography examination in%. Values above 85% will be classified as good sleep efficiency, and values below 85% will be classified as poor sleep efficiency. These polysomnographic exams were performed at the "Sleep Institute of Pelotas (ISP)" from January 2012 to July 2018.
Tabulation of polysomnographic report related to sleep bruxism | The deadline is until May 2020 to have all data collected
  These data are provided from the medical report generated in the polysomnography examination in the presence or absence of sleep bruxism. These polysomnographic exams were performed at the "Sleep Institute of Pelotas (ISP)" from January 2012 to July 2018.
Tabulation of polysomnographic report related to obstructive sleep apnea syndrome (SAOS) | The deadline is until May 2020 to have all data collected
  OSAS is classified according to its severity, which varies according to the number of apnea and hypopnea indexes per hour (AHI), 15; moderate of 16-30, and recorded the first upper 31 episodes. These data are provided from the medical report generated in the polysomnography. These polysomnographic exams were performed at the "Sleep Institute of Pelotas (ISP)" from January 2012 to July 2018.

CONTACTS AND LOCATIONS:
Overall Officials: Noéli Boscato, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil